CLINICAL TRIAL: NCT05011812
Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PBI-0451 in Healthy Subjects.
Brief Title: Study of PBI-0451 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pardes Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBI-0451-0001
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — PBI-0451; Ritonavir; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Open to Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part 1, Treatment A (Experimental): Dose level 1 of PBI-0451
  Interventions: Drug: PBI-0451 Dose 1; Drug: Placebo
- Part 1, Treatment B (Experimental): Dose level 2 of PBI-0451
  Interventions: Drug: PBI-0451 Dose 2; Drug: Placebo
- Part 1, Treatment C (Experimental): Dose level 3 of PBI-0451
  Interventions: Drug: PBI-0451 Dose 3; Drug: Placebo
- Part 1, Treatment D (Experimental): Dose level 4 of PBI-0451
  Interventions: Drug: PBI-0451 Dose 4; Drug: Placebo
- Part 2, Treatment E (Experimental): PBI-0451 =/< Dose level 1
  Interventions: Drug: PBI-0451 Dose 1; Drug: Placebo
- Part 2, Treatment F (Experimental): PBI-0451 =/< Dose level 2
  Interventions: Drug: PBI-0451 Dose 2; Drug: Placebo
- Part 2, Treatment G (Experimental): PBI-0451 =/< Dose level 3
  Interventions: Drug: PBI-0451 Dose 3; Drug: Placebo
- Part 2, Treatment H (Experimental): PBI-0451 =/< Dose level 4
  Interventions: Drug: PBI-0451 Dose 4; Drug: Placebo
- Part 3, Treatment J (Experimental): PBI-0451 + ritonavir (a CYP450 3A inhibitor)
  Interventions: Drug: Ritonavir; Drug: Placebo; Drug: PBI-0451
- Part 3, Treatment K (Experimental): PBI-0451 + ritonavir
  Interventions: Drug: Ritonavir; Drug: Placebo; Drug: PBI-0451
- Part 3, Treatment L (Experimental): PBI-0451 dose TBD
  + midazolam (a sensitive CYP450 3A substrate)
  Interventions: Drug: Midazolam; Drug: Placebo; Drug: PBI-0451
- Part 1, Treatment M (Experimental): Dose level 2 of PBI-0451 with food
  Interventions: Drug: PBI-0451 Dose 2; Drug: Placebo
- Part 2, Treatment I (Experimental): PBI-0451 =/< Dose level 5
  Interventions: Drug: Placebo; Drug: PBI-0451 Dose 5
- Part 1, Treatment N (Experimental): Dose Level 5 of PBI-0451
  Interventions: Drug: Placebo; Drug: PBI-0451 Dose 5

INTERVENTIONS:
Drug: PBI-0451 Dose 1 — Dose level 1 of PBI-0451
  Other Names: PBI-0451
  Arms: Part 1, Treatment A; Part 2, Treatment E
Drug: PBI-0451 Dose 2 — Dose level 2 of PBI-0451
  Other Names: PBI-0451
  Arms: Part 1, Treatment B; Part 1, Treatment M; Part 2, Treatment F
Drug: PBI-0451 Dose 3 — Dose level 3 of PBI-0451
  Other Names: PBI-0451
  Arms: Part 1, Treatment C; Part 2, Treatment G
Drug: PBI-0451 Dose 4 — Dose level 4 of PBI-0451
  Other Names: PBI-0451
  Arms: Part 1, Treatment D; Part 2, Treatment H
Drug: Ritonavir — Ritonavir will be co-administered with the study drug in Treatments J and K
  Other Names: Norvir
  Arms: Part 3, Treatment J; Part 3, Treatment K
Drug: Midazolam — Midazolam will be co-administered with the study drug in Treatment L
  Arms: Part 3, Treatment L
Drug: Placebo — Placebo to match
Drug: PBI-0451 — Dose level of PBI-0451 with a projected exposure
  Arms: Part 3, Treatment J; Part 3, Treatment K; Part 3, Treatment L
Drug: PBI-0451 Dose 5 — Dose level 5 of PBI-0451
  Other Names: PBi-0451
  Arms: Part 1, Treatment N; Part 2, Treatment I

SUMMARY:
This is a phase 1, placebo-controlled, blinded, randomized, dose escalation study of PBI-0451 in healthy subjects. PBI-0451 is a new chemical entity and inhibitor of the main protease of coronaviruses, including the SARS-CoV-2 that causes COVID-19 disease. The study is designed to evaluate the safety, tolerability and pharmacokinetics of PBI-0451 after single and multiple ascending doses and also to explore drug-drug interaction potential of PBI-0451.

DETAILED DESCRIPTION:
Combined Three part, double blind, (sponsor open) study. Part 1: Single ascending dose study. Part 2: Multiple ascending dose study. Part 3: Drug-drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy male or female subjects aged 18-59 years.
2. Body Mass Index (BMI) of ≥ 19.0 and ≤ 30.0 kg/m2.
3. 12-Lead electrocardiogram (ECG) evaluation without clinically significant abnormalities.
4. Normal renal function, including having a creatinine clearance (CLcr) ≥90mL/min
5. Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
6. Screening laboratory assessments must be without clinically significant abnormalities as assessed by the investigator.

Exclusion Criteria:

1. Pregnant and lactating females
2. Have received any investigational drug (or vaccine) within the last 30 days prior to study dosing.
3. Have a positive test result for HIV or HBsAg.
4. Have poor venous access that limits phlebotomy
5. Have taken any prescription medications or over-the-counter medications, including herbal products and dietary supplements within 28 days prior to start of study.
6. Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to Screening or is expected to receive these agents during the study.
7. Have a history of lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
8. Have a history of significant drug sensitivity, cardiac disease, syncope, palpitations, or unexplained dizziness, implanted defibrillator or pacemaker, liver disease, severe peptic ulcer disease, gastroesophageal reflux disease and a medical or surgical treatment that permanently altered gastric absorption.
9. Have received inactivated vaccinations within 4 weeks prior to randomization or receive live vaccinations within 4 weeks of Screening.
10. Received the COVID-19 vaccine either within 7 days or have not completed the series of required 2 doses.
11. Have a history of excessive alcohol use or other illicit drug use within 6 months of screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) in Single Ascending Dose (SAD) compared to placebo | Day 1- Day 14 (From start of study medication till 14 days of last administration of study drug)
  An adverse event is any untoward medical occurrence in patient or clinical study participant temporarily associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect. AEs include both SAEs and AEs. TAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment.
Number of subjects with clinically significant change from Baseline in vital signs in SAD | Day 1-Day 14 (From start of study medication till 14 days of last administration of study drug)
  Vital signs include blood pressure, heart rate, respiratory rate, and temperature
Number of patients with laboratory abnormalities in SAD | Day 1-Day 14 (From start of study medication till 14 days of last administration of study drug)
  Hematology and serum chemistry
Number of subjects with treatment emergent adverse events (TEAEs) in Multiple Ascending Dose (MAD) compared to placebo | Day 1-Day 11, and Follow up (after 14 days)
  An adverse event is any untoward medical occurrence in patient or clinical study participant temporarily associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect. AEs include both SAEs and AEs. TAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment.
Number of subjects with clinically significant change from Baseline in vital signs in MAD | Day 1-Day 11, and Follow up (after 14 days)
  Vital signs include blood pressure, heart rate, respiratory rate, and temperature
Number of patients with laboratory abnormalities in MAD | Day 1-Day 11, and Follow up (after 14 days)
  Hematology and serum chemistry

SECONDARY OUTCOMES:
To collect ECG data for PBI-0451 for the purpose of concentration-QT/QTc modeling | Day 1, 4, 6 and 11
  Criteria for clinically significant changes in ECG (12 lead) are defined as: a postdose QTc interval increase by =/>30msec from the baseline and is >450 msec; or an absolute QTc value is =/> 500 msec for any scheduled ECG.
Plasma concentration of each dose of study drug to determine AUCinf in SAD | Day 1-Day 6
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time 0 to extrapolated infinite time.
Plasma concentration of each dose of study drug to determine AUClast in SAD | Day 1-Day 6
  AUClast is summarized by dosing regimen and determined by linear/log trapezoidal method.
Plasma concentration of each dose of study drug to determine %AUCexp in SAD | Day 1-Day 6
  %AUCexp is summarized by dosing regimen and expressed as area under the plasma concentration-time curve extrapolated from time (tau) to infinity as a percentage of total AUC
Plasma concentration of each dose of study drug to determine CL/F in SAD | Day 1-Day 6
  CL/F is a measure of the rate at which a drug is metabolized or eliminated by normal biological process
Plasma concentration of each dose of study drug to determine CLss/F in MAD | Day 4, Day 6, Day 8
  CLss/F is the total body clearance for extravascular administration divided by the fraction of dose absorbed
Plasma concentration of each dose of study drug to determine AUCtau in MAD | Day 4, Day 6, Day 8
  Area under the plasma concentration- Time profile from Time zero to end of dosing interval. AUCtau is summarized by dosing regimen and period.
Plasma concentration of each dose of study drug to determine Cmax in MAD | Day 4, Day 6, Day 8 (Pre dose to 24 hours)
  Observed Cmax is estimated based on the plasma concentrations.
Plasma concentration of each dose of study drug to determine Tmax in MAD | Day 4, Day 6, Day 8 (Pre dose to 24 hours)
  Tmax is summarized by dosing regimen
Plasma concentration of each dose of study drug to determine Tlast in MAD | Day 4, Day 6, Day 8
  Tlast is the time of last measurable concentration
Plasma concentration of each dose of study drug to determine Clast in MAD | Day 4, Day 6, Day 8
  Clast is the last measurable concentration (above the quantification limit)
Plasma concentration of each dose of study drug to determine Ctau in MAD | Day 4, Day 6, Day 8
  Ctau is the concentration at the end of dosing interval
Plasma concentration of each dose of study drug to determine λz in MAD | Day 4, Day 6, Day 8
  Individual estimate of terminal elimination rate constant, calculated using log-linear regression of the terminal portions of the plasma concentration-versus-time curves.
Plasma concentration of each dose of study drug to determine t1/2 | Day 1(0 hours- 24 hours post dose), Day 4, Day 6, Day 8
  t1/2 is summarized by dosing regimen . It is determined by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline is used in the regression.
Plasma concentration of each dose of study drug to determine Vz/F | Day 4, Day 6, Day 8
  Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. VZ/F after oral dose is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Marshall, Principal Investigator — New Zealand Clinical Research
Locations (1):
- Auckland City Hospital, Auckland, New Zealand